CLINICAL TRIAL: NCT04954339
Title: DYNAmic Immune Microenvironment of HCC Treated With atezolIzumab Plus bevaCizumab
Acronym: DYNAMIC
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tae Won Kim (Other)
Responsible Party: Sponsor-Investigator, Tae Won Kim, PhD, Asan Medical Center
Organization: Asan Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-0785
Record Dates: First submitted 2021-06-08; First posted 2021-07-08 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Atezolizumab plus Bevacizumab (Experimental): Two cycles of naeoadjuvant atezolizumab (1200 mg) plus bevacizumab (15 mg/kg) prior to surgical resection and four cycles of adjuvant atezolizumab (1200 mg) plus bevacizumab (15 mg/kg) after the surgery will be administered.
  Interventions: Drug: Aatezolizumab plus Bevacizumab

INTERVENTIONS:
Drug: Aatezolizumab plus Bevacizumab — Two cycles of naeoadjuvant atezolizumab (1200 mg) plus bevacizumab (15 mg/kg) prior to surgical resection and four cycles of adjuvant atezolizumab (1200 mg) plus bevacizumab (15 mg/kg) after the surgery will be administered.
  Other Names: Ticentriq plus Avastin

SUMMARY:
Part I (Clinical trial setting): A single-arm phase II study to investigate the efficacy of neoadjuvant atezolizumab (T) + bevacizumab (A) in patients with potentially resectable BCLC stage B/C or high risk resectable hepatocellular carcinoma (HCC) (n = 45)

Part II (Biomarker study setting): Exploratory translational research will be conducted using samples obtained from Part 1 (n =45) and those acquired from an independent cohort of treatment-naïve HCC patients (n = 15).

DETAILED DESCRIPTION:
Same as above

ELIGIBILITY:
Inclusion Criteria:

* Acquisition of Signed Informed Consent Form prior to any study specific procedures
* Willingness and ability to comply with the study protocol
* ≥ 19 years of age at the time of signing Informed Consent Form
* Eastern Cooperative Oncology Group (ECOG) performance status of ≤1
* Histologically or cytologically confirmed HCC
* Child-Pugh class A (Child-Pugh score of 5 or 6) assessed within 7 days
* Negative HIV test at screening
* Documented virology status of hepatitis, as confirmed by screening HBV and HCV serology test
* For patients with active hepatitis B virus (HBV): HBV DNA < 500 IU/mL obtained within 28 days prior to initiation of study treatment, and Anti-HBV treatment (per local standard of care; e.g., entecavir) for a minimum of 14 days prior to study entry and willingness to continue treatment for the length of the study
* Potentially resectable Barcelona Clinic Liver Cancer (BCLC) stage B/C meeting any of the following criteria by 4-phase liver dynamic computed tomography (CT) or gadoxetic-acid enhanced magnetic resonance imaging (MRI) or chest CT with enhancement
* Portal vein invasion (Vp1, Vp2 and Vp3)
* Hepatic vein invasion (Vv1 and Vv2)
* Lymph node metastasis
* multiple tumor nodules (n ≥ 2)
* Solitary distant metastasis or Resectable HCC meeting any of the following criteria by 4-phase liver dynamic CT or gadoxetic-acid enhanced MRI
* Serum alpha-feto protein (AFP) level of ≥ 400ng/mL
* Largest tumor diameter of ≥ 5cm
* Presence of satellite nodules
* Presence of ≥ 1 measurable untreated lesion (per RECIST v1.1)
* One or more hepatic lesions should be accessible for biopsy
* Adequate major organ functions as following:
* Hematopoietic function: absolute neutrophil count (ANC) ≥ 1,500/mm3, Platelet ≥ 75,000/mm3
* Hemoglobin ≥ 90 g/L (9 g/dL). Patients may be transfused to meet this criterion.
* Serum albumin ≥ 28 g/L (2.8 g/dL) without transfusion
* Hepatic function: serum bilirubin 2 x ULN, AST/ALT levels 5 x ULN
* Renal function: serum creatinine 1.5 x ULN or creatinine clearance ≥ 50 mL/min (calculated using
* the Cockcroft-Gault formula)
* PT INR < 1.5 or aPTT < 1.5 x ULN within 14 days prior to the start of study treatment for patients not receiving anti-coagulation. For patients receiving anticoagulants, INR and aPTT must be within the medical standard of enrolling institution.
* For women of childbearing potential

Exclusion Criteria:

* Extrahepatic metastases that are not candidates for treatment of curative aim (e.g. resection, radiation or radiofrequency ablation)
* Presence of central nervous system (CNS) metastases
* Concurrent or previous history of another primary cancer within 3 years prior to study treatment except for curatively treated cervical cancer in situ, non-melanomatous skin cancer, superficial bladder cancer (pTis or pT1) and curatively treated thyroid cancer of any stage. Concurrent, histologically confirmed, unresected thyroid cancer without distant metastasis could be allowed with the agreement of the principal investigator.
* Chronic hepatitis B, defined as HBV DNA (> 2,000 IU / mL) and ALT> upper limit of normal range, must be treated with antiviral drugs before enrollment to reach appropriate viral suppression (HBV DNA <2000 IU / mL), and the antiviral drugs must be maintained during the study treatment period and for 6 months after the last dose of study treatment.
* Prior systemic therapy for metastatic disease including systemic investigational agents
* Uncontrolled medical illness: including medically uncontrolled infection, uncontrolled hypertension, unstable angina, symptomatic congestive heart failure, myocardial infarction within 6 months
* Current or recent (within 10 days of start of study treatment) use of aspirin (>325mg/day), clopidogrel (>75mg/day), oral or parenteral anticoagulants or thrombolytic agents for therapeutic purposes (therapeutic anticoagulation on a stable dose for at least 2 weeks prior to the start of study treatment is allowed)
* Known alcohol or drug abuse- Severe infection within 4 weeks prior to initiation of study treatment, including, but not limited to, hospitalization for complications of infection, bacteremia, or severe pneumonia
* Treatment with therapeutic oral or IV antibiotics within 2 weeks prior to initiation of study treatment.
* Patients receiving prophylactic antibiotics (e.g., to prevent a urinary tract infection or chronic obstructive pulmonary disease exacerbation) are eligible for the study.
* Inadequately controlled hypertension (defined as systolic blood pressure >150mmHg and/or diastolic blood pressure >100mmHg)
* Prior history of hypertensive crisis or hypertensive encephalopathy
* History or evidence upon physical or neurological examination of CNS disease (e.g. seizures) unrelated to cancer unless adequately treated with standard medical therapy
* Significant vascular disease (e.g. aortic aneurysm requiring surgical repair or recent arterial thrombosis) within 6 months of start of study treatment
* Significant cardiovascular disease (such as New York Heart Association Class II or greater cardiac disease, myocardial infarction, or cerebrovascular accident within 3 months prior to initiation of study treatment), unstable arrhythmia, or unstable anginanginaa
* Major surgical procedure, other than for diagnosis, within 4 weeks prior to initiation of study treatment, or anticipation of need for a major surgical procedure during the study
* History of congenital long QT syndrome or corrected QT interval > 500 ms (calculated with use of Fridericia method) at screening
* History of uncorrectable electrolyte disorder affecting serum levels of potassium, calcium, magnesium
* Any previous venous thromboembolism > CTCAE Grade 3 within 12 months prior to start of study treatment
* History of hemoptysis (≥ 2.5 mL of bright red blood per episode) within 1 month prior to initiation of study treatment
* Any previous venous thromboembolism > CTCAE Grade 3 within 12 months prior to start of study treatment
* History of abdominal fistula, gastrointestinal perforation, intra-abdominal abscess or active GI bleeding within 6 months prior to start of study treatment
* Serious, non-healing wound, active ulcer, or untreated bone fracture
* Known hypersensitivity to any component of any of the study medication
* History of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanised antibodies or fusion proteins
* Pregnant or breastfeeding, or intending to become pregnant during the study or within 6 months after the last dose of study treatment
* Positive serum or urine pregnancy test: Women of childbearing potential must have a negative serum or urine pregnancy test result within 14 days prior to initiation of study treatment to be enrolled to this study.
* Known hypersensitivity or allergy to Chinese hamster ovary cell products
* Active or history of autoimmune disease or immune deficiency, including, but not limited to, myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, antiphospholipid antibody syndrome, Wegener granulomatosis, Sjögren's syndrome, Guillain-Barré syndrome, or multiple sclerosis, with the following exceptions:

Patients with a history of autoimmune-related hypothyroidism who are on thyroid replacement hormone are eligible for the study.

Patients with controlled Type 1 diabetes mellitus who are on an insulin regimen are eligible for the study.

Patients with eczema, psoriasis, lichen simplex chronical, or vitiligo with dermatologic manifestations only (e.g., patients with psoriatic arthritis are excluded) are eligible for the study provided all of following conditions are met:

Rash must cover < 10% of body surface area Disease is well controlled at baseline and requires only low-potency topical corticosteroids No occurrence of acute exacerbations of the underlying condition requiring psoralen plus ultraviolet A radiation, methotrexate, retinoids, biologic agents, oral calcineurin inhibitors, or high potency or oral corticosteroids within the previous 12 months

* Prior allogeneic bone marrow transplantation or prior solid organ transplantation
* History of idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, or idiopathic pneumonitis, or evidence of active pneumonitis on screening chest computed tomography (CT) scan History of radiation pneumonitis in the radiation field (fibrosis) is permitted.
* A prior bleeding event due to esophageal and/or gastric varices within 6 months prior to initiation of study treatment
* Positive test for human immunodeficiency virus (HIV)
* Co-infection of HBV and HCV Patients with a history of HCV infection but who are negative for HCV RNA by PCR will be considered non-infected with HCV.
* Active tuberculosis
* Administration of a live, attenuated vaccine within 4 weeks prior to start of study treatment or anticipation that such a live attenuated vaccine will be required during the study
* Prior treatment with CD137 agonists, anti-CTLA4, anti-PD-1, or anti-PD-L1 therapeutic antibody or pathway-targeting agents
* Treatment with systemic immunostimulatory agents
* Treatment with systemic corticosteroids or other systemic immunosuppressive medications

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-10-29 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The rate of major pathological response | Through treatment discontinuation, an average of 6 months
  Part I_The rate of major pathological response (MPR) rate defined by <10% of residual viable tumor in the tumor bed
Distinct immunophenotypes and dynamic changes of tumor-infiltrating immune cells by single nucelar RNA-sequencing, single cell RNA sequencing, spatial transcriptomics, multiplexed immunohistochemistry (mIHC), flow cytometry (and/or CyTOF) | up to 36 months
  Part II_Rate of single nucelar RNA-sequencing, single cell RNA sequencing, spatial transcriptomics, multiplexed immunohistochemistry (mIHC), flow cytometry (and/or CyTOF)

SECONDARY OUTCOMES:
The rate of completion of treatment and resection | Through treatment discontinuation, an average of 6 months
  Part I_The rate of completion of treatment is defined by the proportion of patients receiving all of the planned treatments
The rate of R0 resection | Through treatment discontinuation, an average of 6 months
  Part I_The rate of resection is defined as the proportion of patients completing 2 cycles of Atezolizumab plus Bevacizumab
Incidence and severity of adverse events, with severity determined according to Common Terminology Criteria for Adverse Events v5.0 | up to 36 months
  Part I_Incidence and severity of adverse events
Progression-free survival (PFS) | up to 36 months
  Part I_Progression free survival
Radiological response | From enrol to surgical resection, an average 6 months
  Part I_Radiological response is determined by the investigator according to the RECIST (Response evaluation criteria in solid tumor) V1.1
Recurrence-free survival (RFS) | Through treatment discontinuation, an average of 6 months
  Part I_Recurrence-free survival (RFS) for those who achieved R0 resection
Distinct immunophenotypes of tumor-infiltrating immune cells of HCCs treated with T+A in comparison with those of treatment-naïve HCCs assessed by multicolor flow cytometry and CyTOF. | up to 36 months
  Part_II
Characterization of immunologic and genomic features | up to 36 months
  Part II_- Single nuclear RNA sequencing (snRNA seq), T-cell receptor (TCR) sequencing, multi-color flow cytometry (and/or cyTOF), multiplexed immunohistochemistry (mIHC) and whole genome sequencing (WGS)
Comparison of immunophenotypes and immune landscapes of tumor-infiltrating immune cells | up to 36 months
  Part II_Comparison of immunophenotypes and immune landscapes of tumor-infiltrating immune cells of atezolizumab-bevacizumab -treated hepatocelluar carcinoma's with those of treatment naïve hepatocelluar carcinoma
Dynamic changes in T-cell receptor (TCR) repertoire of peripheral mononuclear cells | up to 36 months
  Part II_Dynamic changes in T-cell receptor (TCR) repertoire of peripheral mononuclear cells following atezolizumab-bevacizumab treatment

CONTACTS AND LOCATIONS:
Overall Officials: Tae Won Kim, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, Songpa, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bray F, Ferlay J, Soerjomataram I, Siegel RL, Torre LA, Jemal A. Global cancer statistics 2018: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2018 Nov;68(6):394-424. doi: 10.3322/caac.21492. Epub 2018 Sep 12. PMID 30207593
- [Background] El-Serag HB. Hepatocellular carcinoma. N Engl J Med. 2011 Sep 22;365(12):1118-27. doi: 10.1056/NEJMra1001683. No abstract available. PMID 21992124
- [Background] Forner A, Llovet JM, Bruix J. Hepatocellular carcinoma. Lancet. 2012 Mar 31;379(9822):1245-55. doi: 10.1016/S0140-6736(11)61347-0. Epub 2012 Feb 20. PMID 22353262
- [Background] Heimbach JK, Kulik LM, Finn RS, Sirlin CB, Abecassis MM, Roberts LR, Zhu AX, Murad MH, Marrero JA. AASLD guidelines for the treatment of hepatocellular carcinoma. Hepatology. 2018 Jan;67(1):358-380. doi: 10.1002/hep.29086. No abstract available. PMID 28130846
- [Background] Chan AWH, Zhong J, Berhane S, Toyoda H, Cucchetti A, Shi K, Tada T, Chong CCN, Xiang BD, Li LQ, Lai PBS, Mazzaferro V, Garcia-Finana M, Kudo M, Kumada T, Roayaie S, Johnson PJ. Development of pre and post-operative models to predict early recurrence of hepatocellular carcinoma after surgical resection. J Hepatol. 2018 Dec;69(6):1284-1293. doi: 10.1016/j.jhep.2018.08.027. Epub 2018 Sep 18. PMID 30236834